CLINICAL TRIAL: NCT03204045
Title: Comparison of the Effects of Oxycodone Versus Fentanyl on Airway Reflex to Tracheal Extubation and Postoperative Pain During Recovery of Anesthesia After Laparoscopic Cholecystectomy
Brief Title: Comparison of the Effects of Oxycodone Versus Fentanyl on Airway Reflex to Tracheal Extubation and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-06-26
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Coughing Responses at Tracheal Extubation
Keywords: oxycodone, fentanyl, tracheal extubation
MeSH Terms: interventions — Fentanyl; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fentanyl (Active Comparator): fentanyl 1 ㎍/kg
  Interventions: Drug: Oxycodone; Drug: control
- oxycodone (Active Comparator): oxycodone 0.08 mg/kg
  Interventions: Drug: fentanyl; Drug: control
- control (Placebo Comparator): isotonic saline
  Interventions: Drug: fentanyl; Drug: Oxycodone

INTERVENTIONS:
Drug: fentanyl — 2 mL mixture of fentanyl with isotonic saline
  Arms: control; oxycodone
Drug: Oxycodone — 2 mL mixture of oxycodone with isotonic saline
  Arms: control; fentanyl
Drug: control — isotonic saline 2 mL
  Arms: fentanyl; oxycodone

SUMMARY:
This study was performed to compare the effects of oxycodone and fentanyl on airway and hemodynamic responses and postoperative pain during recovery period in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This study was approved by the committee of Institutional Review Board of the Yeungnam University Hospital, Daegu, Republic of Korea. 90 patients were enrolled in this study and written informed consent was obtained from all patients. We included patients with ASA physical status classification I or II, and aged 18-65 years scheduled for elective laparoscopic cholecystectomy.

Patients were assigned to one of three groups by computer-generated randomization, fentanyl group (group F, N=30), oxydodone group (group O, N=30), or control group (group C, N=30). 10 minutes before completion of surgery, patients received 2 mL mixture of fentanyl 1 ㎍/kg or oxycodone 0.08 mg/kg with isotonic saline or isotonic saline 2 mL intravenously in accordance with allocated study groups by an anesthesiologist who was blinded to group treatment.

Airway reflex responses including coughing, breath holding, bucking, and laryngospasm were recorded at point of awareness, extubation, and 3 min after tracheal extubation. Hemodynamic responses were recorded at the completion of surgery (T1), at the point of awareness (T2), at the point of extubation (T3), and 3 min after tracheal extubation (T4). Coughing severity was assessed using a 5-point scale. In the recovery room, hemodynamic responses were evaluated every 5 min for 30 min. The postoperative pain intensity was assessed 5 and 30 min in the postanesthetic care unit (PACU) using numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification I or II, and aged 18-65 years scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* allergy to either fentanyl or oxycodone, history of chronic other opioids or analgesics use, history of cardiac, hepatic, or renal disease, other comorbid conditions, cognitive impairment or body mass index more than 35 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
airway response | at point of awareness (eye opening in response to verbal commands), extubation, and 3 min after tracheal extubation
  incidence of coughinging
postoperative pain | 5 and 30 min in the postanesthetic care unit
  numerical rating scale ranging from 0 (no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, Nam-gu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes